CLINICAL TRIAL: NCT06175845
Title: Radiofrequency Ablation Via Catheter and Transpapillary Access in Patients With Cholangiocarcinoma
Brief Title: Endoscopic Radiofrequency Ablation for Unresectable Cholangiocarcinoma
Acronym: ACTICCA-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johann von Felden, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0645/131
Record Dates: First submitted 2023-11-25; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cholangiocarcinoma; Klatskin Tumor; Bile Duct Cancer; Liver Cancer
Keywords: Radiofrequency ablation; Intraductal; Biliary; Endoscopic retrograde cholangiography; Transpapillary; Stent dysfunction; Cholangitis; Obstruction
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Bile Duct Neoplasms; Liver Neoplasms; Cholangitis; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: ablation arm (Active Comparator): Systemic chemotherapy and bile duct stenting with intraductal RFA of malignant bile duct obstructions employing a CE-certified ablation catheter prior to stent placement.
  Interventions: Procedure: Intraductal biliary radiofrequency ablation
- Arm B: control arm (No Intervention): Systemic chemotherapy and bile duct stenting without RFA.

INTERVENTIONS:
Procedure: Intraductal biliary radiofrequency ablation — Radiofrequency ablation via catheter and transpapillary access of malignant bile duct obstruction
  Other Names: RFA
  Arms: Arm A: ablation arm

SUMMARY:
The goal of this clinical trial is to learn about radiofrequency ablation in patients with unresectable bile duct cancer who receive systemic chemotherapy and bile duct stenting. The main questions it aims to answer are:

* Does radiofrequency ablation of tumorous bile duct occlusion reduce risk of complications in these patients (eg stent dysfunction, delay of chemotherapy, infections etc)?
* Is radiofrequency ablation safe in these patients? All participants will receive standard treatment with systemic chemotherapy and bile duct stenting. Researchers will compare two groups (one group will receive additional radiofrequency ablation, the other not).

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable perihilar and/or ductal CCA with bile duct stenting and palliative systemic therapy as indicated by the local Multidisciplinary Team (MDT)
2. Written informed consent
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Age ≥18 years
5. Eligibility for palliative systemic therapy based on clinical and laboratory parameters (except hyperbilirubinemia) as determined by the local MDT
6. No prior radiofrequency ablation (RFA) for CCA
7. No repeated bile duct stenting in the past 3 months (trial inclusion is possible upon first stent replacement or initial stent placement within past 3 months)
8. No concomitant disease or malignancy interfering with the study procedure or efficacy outcome measures, particularly no severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, myocardial infarction within ≤3 months, significant arrhythmias) and no psychiatric disorders precluding understanding of information of trial related topics and giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time to first event, ie stent dysfunction | 6 months
  • Time-to-first event (during 6 months follow up), i.e. stent dysfunction defined by bilirubin >5 mg/dl and/or cholangitis (fever >38.5°C and/or increase in C-reactive protein by at least 3-fold upper limit of normal and at least 20% from baseline without extrahepatic focus and absence of tumor progression) leading to premature stent replacement and/or disruption of chemotherapy (all possible events will be reviewed by a blinded and independent Endpoint Review Committee [ERC].)

SECONDARY OUTCOMES:
Overall survival | up to 30 month
  Time to death or last seen alive
Satisfaction assessed by EORTC QLQ-C30 questionnaire | 6 months
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in cancer patients. It is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Satisfaction assessed by EORTC QLQ-BIL21 questionnaire | 6 months
  The EORTC QLQ-BIL21 consists of 21 questions: 3 single-item assessments relating to treatment side effects, difficulties with drainage bags/tubes and concerns regarding weight loss, in addition to 18 items grouped into 5 proposed scales: eating symptoms (4 items), jaundice symptoms (3 items), tiredness (3 items), pain symptoms (4 items) and anxiety symptoms (4 items). The response format is a four-point Likert scale.and designed to more specifically adress side effects.
  A high scale score represents a higher response level.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE V5 | 6 months
  Safety events
Clinical event rate at 6 months | 6 months
  Rate of clinical events defined as per primary outcome after 6 months follow up
Total days of overnight-hospital-stays | 6 months
  Total days of overnight-hospital-stays

CONTACTS AND LOCATIONS:
Overall Officials: Johann von Felden, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Schmidt C, Zapf A, Ozga AK, Canbay A, Denzer U, De Toni EN, Lohse AW, Schulze K, Rosch T, Stein A, Wege H, von Felden J. Radiofrequency ablation via catheter and transpapillary access in patients with cholangiocarcinoma (ACTICCA-2 trial) - a multicenter, randomized, controlled, open-label investigator-initiated trial. BMC Cancer. 2024 Aug 1;24(1):931. doi: 10.1186/s12885-024-12693-w. PMID 39090600